CLINICAL TRIAL: NCT00286104
Title: The Impact of Ventricular Catheter Impregnated With Antimicrobial Agents on Infection in Patients With Ventricular Catheter: A Prospective Randomized Study
Brief Title: Impact of Ventricular Catheter Used With Antimicrobial Agents on Patients With a Ventricular Catheter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: George KC Wong, Division of Neurosurgery, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CREC-PWS-002
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-07

CONDITIONS: Hydrocephalus; Intracranial Hypertension
Keywords: Ventriculitis; External ventricular catheter; Antibiotic-impregnated
MeSH Terms: conditions — Hydrocephalus; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bactiseal ventricular catheter (Rifampicin- and Clindamycin-impregnated)
  Interventions: Device: Antibiotics-impregnated ventricular catheter (Bactiseal®)
- 2 (Placebo Comparator): Plain ventricular catheter
  Interventions: Device: Plain ventricular catheter (Codman EDS II/III)

INTERVENTIONS:
Device: Antibiotics-impregnated ventricular catheter (Bactiseal®) — Antibiotics-impregnated ventricular catheter (Rifampicin- and Clindamycin-impregnated)
  Other Names: Bactiseal
  Arms: 1
Device: Plain ventricular catheter (Codman EDS II/III) — Plain ventricular catheter
  Other Names: Codman EDS II/III
  Arms: 2

SUMMARY:
External ventricular catheters are used for intracranial pressure monitoring and temporary cerebrospinal fluid (CSF) drainage in neurosurgery. The incidence of ventriculostomy-related cerebrospinal fluid infections had been quoted as between 2.2% to 10.4% in the more recent literature. Previous prospective studies in the investigators' unit have shown that the use of dual antibiotics prophylaxis in patients with external ventricular drain was associated with decreased incidence of CSF infection but was complicated with opportunistic extracranial infections. The current practice is to cover with prophylactic dual antibiotics unless guided by microbiology results for all patients with external ventricular drain. In recent years, cerebrospinal fluid shunt catheters impregnated with antimicrobial agents have been available. Experimental studies have shown that they provide protection against staphylococcal aureus and coagulase-negative staphylococci strains for between 42 days and 56 days. Theoretically, they provide the antibiotic prophylaxis locally without the associated complications of systemic antibiotics.

It is hypothesized that the use of antibiotic-impregnated catheters instead of systemic antibiotic prophylaxis will not increase the rate of cerebrospinal fluid infection, will decrease the rate of opportunistic/nosocomial infections and improves the overall outcome in these patients; that would convert into a reduction in treatment cost of these patients.

DETAILED DESCRIPTION:
Objective:

1. To assess the cranial and extracranial infection rate of systemic antibiotic prophylaxis versus antibiotics-impregnated catheter.
2. To assess the patients' outcome and carry out cost analysis for systemic antibiotic prophylaxis versus antibiotics-impregnated catheter.

Design: Prospective randomized controlled trial

Hypothesis: The use of antibiotics-impregnated catheter instead of systemic antibiotic prophylaxis will not increase the rate of cerebrospinal fluid infection, will decrease the rate of opportunistic/nosocomial infection and improves the overall outcome in these patients; that would convert into a reduction in treatment cost of these patients.

Method: After ventricular catheter insertion, patients will be randomized into one of the two groups:

1. Periprocedural antibiotics: Only ie Unasyn and Rocephin and insertion of the antibiotics-impregnated ventricular catheter.
2. Periprocedural antibiotics and prophylactic dual antibiotics ie Unasyn and Rocephin and insertion of ventricular catheter without impregnation of antibiotics.

Primary outcome variable: Cerebrospinal fluid infection and extracranial infection.

Sample size: We aim to recruit a total of 180 patients with 90 patients in each arm and expect to complete patient recruitment in 2-3 years. The calculation is based to detect a difference of nosocomial infection rate between 20% and 40%, with 5% level of significance and 80% power.

Projected results and significance:

The project has a good chance to be the first clinical study to the outcome and cost impacts of antibiotic-impregnated ventricular catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with external ventricular drain inserted
2. Patients with external ventricular drain in-situ planned for at least 5 days

Exclusion Criteria:

1. Known CSF infection including meningitis
2. Known sepsis
3. Uncorrected coagulopathy
4. No consent available

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2004-04; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid infection rate | First 30 days
Extracranial infection rate | First 30 days

SECONDARY OUTCOMES:
Mortality rate | At discharge and six months
Glasgow Outcome Scale Extended | At discharge and at six months

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, FRCSEd(SN), Principal Investigator — Chinese University of Hong Kong; George KC Wong, FRCSEd(SN), Study Director — Chinese University of Hong Kong
Locations (1):
- Division of Neurosurgery, Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Wong GK, Ip M, Poon WS, Mak CW, Ng RY. Antibiotics-impregnated ventricular catheter versus systemic antibiotics for prevention of nosocomial CSF and non-CSF infections: a prospective randomised clinical trial. J Neurol Neurosurg Psychiatry. 2010 Oct;81(10):1064-7. doi: 10.1136/jnnp.2009.198523. Epub 2010 May 12. PMID 20466698